CLINICAL TRIAL: NCT02881190
Title: A Tolerance, Safety and Pharmacokinetic Ascending Dose Phase I Study of RC48-ADC Administered Intravenously to Subjects With HER2-Positive Malignant in Advanced Malignant Solid Tumors
Brief Title: Study of RC48-ADC Administered Intravenously to Subjects With HER2-Positive in Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C002 CANCER
Record Dates: First submitted 2016-08-20; First posted 2016-08-26 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC (Experimental): The phase I component has several dose levels of RC48-ADC (0.1mg/kg，0.5 mg/kg, 1.0mg/kg, 1.5mg/kg, 2.0mg/kg, 2.5mg/kg, 3.0mg/kg, 3.5mg/kg and 4.0 mg/kg) and is designed as a traditional dose-escalation study.Dosing interval is once two weeks.
  Interventions: Drug: RC48-ADC

INTERVENTIONS:
Drug: RC48-ADC

SUMMARY:
A tolerance, safety and pharmacokinetic ascending dose phase I Study of RC48-ADC administered intravenously to subjects with HER2-positive malignant in advanced malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Aged 18-75 years;
* ECOG physical condition is 0 or 1;
* Life expectancy greater than 12 weeks;
* Patients with locally advanced or metastatic malignant solid tumors diagnosed by pathology and refractory to standard of care therapy, or for whom no standard of care therapy is available histology standard of care therapy, or for whom no standard of care therapy is available;
* Human epidermal growth factor receptor 2 (HER2)-positive refers to immunohistochemistry (IHC 2+or 3+);
* Patients with measurable and appreciable tumor lesions according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1);
* Adequate organ function as defined by the following criteria:

  * absolute neutrophil count(ANC) >= 1.5 x 10(9)/L;
  * platelets>=100*10(9)/L;
  * Total serum bilirubin <=1.5*ULN;
  * serum aspartate transaminase (AST) and serum alanine transaminase (ALT) <=3.0*upper limit of normal (ULN), or AST and ALT<=5*ULN if liver function abnormalities are due to underlying malignancy;
  * normal serum creatinine;
  * international normalized ratio(INR) and activated partial thromboplastin time (aPTT) must be less than or equal to 1.5 times the upper limit of the normal range (ULN);
* Women of child-bearing potential and men must agree to use adequate contraception (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], complete sexual abstinence, or sterilized partner) prior to study entry and during the period of therapy and for 30 days after the last dose of study drug;
* Left ventricular ejection fraction (LVEF) >= 50% as assessed by echocardiogram.

Exclusion Criteria:

* Current pregnancy or lactation;
* Serologic status reflecting active hepatitis B or C infection;
* Major surgery within 4 weeks of first dose of study drug and not fully recovered
* Receiving palliative radiation therapy for bone metastases if administered <= 2 weeks prior to first study treatment;
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4), grade less than or equal to1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia;
* Prior-treatment with other clinical research anticancer drugs within 28 days before study drug treatment;
* The active infection with clinical significance According to the researcher's judgment,
* Known history of immune deficiency,including HIV-positive or other known acquired or congenital immunodeficiency, or organ transplantation;
* Currently active clinically significant cardiovascular disease such as uncontrolled arrhythmia, congestive heart failure, or greater than or equal to Class 2 congestive heart failure as defined by the New York Heart Association Functional Classification, or history of myocardial infarction unstable angina, or acute coronary syndrome within 6 months prior to enrollment in the study;
* Unwilling or unable to participate in all required study evaluations and procedures;
* The time interval which is from the last chemotherapy or HER2 targeted therapy until the first trial is more than 21 days;
* Patients who had received systemic steroid therapy for a long time (Patients who had received systemic steroid therapy for short time and stopped drug more than 2 weeks could be enrolled);
* Serious complications such as active alimentary tract hemorrhage, intestinal obstruction, enteroparalysis, interstitial pneumonia, pulmonary fibrosis, renal failure, glaucoma and uncontrolled diabetes;
* Uncontrolled primary or metastatic tumor of brain;
* Current peripheral neuropathy of Grade ≥ 2;
* History of nerve or psychiatric disorders.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2015-12-14 (Actual); Primary Completion 2019-06-27 (Actual); Study Completion 2019-11-08 (Actual)

PRIMARY OUTCOMES:
Maximal Tolerance Dose (MTD) of RC48-ADC | DLT will be evaluated on Day 28 during cycle 1
  The dose level in which >= 2 out of 6 patients have dose-limiting toxicity (DLT). The MTD is defined as the previous dose level.

SECONDARY OUTCOMES:
Safety (the drug safety as assessed by NCI-CTCAE v4.0) | up to 2 years
  The drug safety as assessed by NCI-CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xu Y, Wang Y, Gong J, Zhang X, Peng Z, Sheng X, Mao C, Fan Q, Bai Y, Ba Y, Jiang D, Yang F, Qi C, Li J, Wang X, Zhou J, Lu M, Cao Y, Yuan J, Liu D, Wang Z, Fang J, Shen L. Phase I study of the recombinant humanized anti-HER2 monoclonal antibody-MMAE conjugate RC48-ADC in patients with HER2-positive advanced solid tumors. Gastric Cancer. 2021 Jul;24(4):913-925. doi: 10.1007/s10120-021-01168-7. Epub 2021 May 4. PMID 33945049